CLINICAL TRIAL: NCT00013182
Title: Effect of Activity on Sleep of Cognitively-Impaired Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: Central Arkansas Veterans Healthcare System (U.S. Federal Agency); University of Arkansas (Other)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: NRM 95-184
Record Dates: First submitted 2001-03-14; First posted 2001-03-16 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2007-02

CONDITIONS: Alzheimer's Disease; Sleep Disorders
MeSH Terms: conditions — Alzheimer Disease; Sleep Wake Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Behavioral: social activity

INTERVENTIONS:
Behavioral: social activity

SUMMARY:
Sleep-activity rhythm disturbance is a prevalent, disabling symptom in cognitively-impaired (CI) elders. Their nocturnal sleep is light and inefficient with frequent awakenings. Multiple short daytime napping episodes interfere with daytime activity and functioning. Daytime disruptive behaviors, such as pacing, hitting, and cursing are related significantly to sleep-activity rhythm disturbance. Medical treatment for sleep and behavior disturbances with benzodiazepines or antipsychotic medications has proven minimally effective and has serious side effects such as impairments in cognition, memory, coordination, and balance, tolerance and severe rebound insomnia, and tardive dyskinesia.

DETAILED DESCRIPTION:
Background:

Sleep-activity rhythm disturbance is a prevalent, disabling symptom in cognitively-impaired (CI) elders. Their nocturnal sleep is light and inefficient with frequent awakenings. Multiple short daytime napping episodes interfere with daytime activity and functioning. Daytime disruptive behaviors, such as pacing, hitting, and cursing are related significantly to sleep-activity rhythm disturbance. Medical treatment for sleep and behavior disturbances with benzodiazepines or antipsychotic medications has proven minimally effective and has serious side effects such as impairments in cognition, memory, coordination, and balance, tolerance and severe rebound insomnia, and tardive dyskinesia.

Objectives:

The degree of daytime sleepiness in elders may reflect a reduction in the purposive physical, cognitive, and affective activities that previously sustained daytime alertness and promoted psychological well-being. For some institutionalized elders, living in a physically, cognitively, and emotionally understimulating setting may induce excessive napping during the day with a subsequent adverse impact on circadian sleep-wake patterns. Concrete, reality-based activities may counter napping by keeping residents with dementia involved in the world around them and helping them meet psychological, physical, and social needs. Our pilot study with five nursing home residents demonstrated that activities timed to occur during usual naptime and tailored to residents� interests and their remaining abilities improved nocturnal sleep. Our other research has shown that engaging residents in meaningful activity improved their psychological well-being and decreased certain types of disruptive behaviors.

Methods:

We tested the effect of an Individualized Activity Intervention timed to occur when the resident usually napped in the daytime on nocturnal sleep as measured by actigraphy in CI nursing home residents. Examples of individualized activities include objects for tactile and visual stimulation, arts and crafts, and games. We also tested the effect of the intervention on psychological well-being and disruptive behavior, and measured its cost. After the collection of baseline sleep, disruptive behavior, and psychological well-being data for five days, residents were randomly assigned to the Individualized Activity Intervention or to a usual care control condition for 21 days. On days 17-21, the research assistant repeated the outcome measures.

Status:

Secondary data analysis on psychological well-being, disruptive behavior, and cost of the intervention is in progress.

ELIGIBILITY:
Inclusion Criteria:

Participants must have been a resident in the nursing home for at least two weeks, must be at least 55 years old, have a diagnosis of dementia, a Mini-Mental State Examination Score of <24, sleep less than 85% of the night, and nap at least 30 minutes during the day.

Exclusion Criteria:

Min Age: 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Study Completion 2001-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen C. Richards, PhD RN, Principal Investigator — Central Arkansas Veterans Healthcare System Eugene J. Towbin Healthcare Center, Little Rock, AR
Locations (1):
- Central Arkansas Veterans Healthcare System Eugene J. Towbin Healthcare Center, Little Rock, AR, No. Little Rock, Arkansas, United States

REFERENCES:
- [Result] Richards KC, Beck C, Shue VM, O'Sullivan PS. Demographic and sleep characteristics in cognitively impaired nursing home residents with and without severe sleep/wake pattern inefficiency. Issues Ment Health Nurs. 2005 Aug-Sep;26(7):751-69. doi: 10.1080/01612840591008339. PMID 16126650
- [Result] Richards KC, Beck C, O'Sullivan PS, Shue VM. Effect of individualized social activity on sleep in nursing home residents with dementia. J Am Geriatr Soc. 2005 Sep;53(9):1510-7. doi: 10.1111/j.1532-5415.2005.53460.x. PMID 16137280
- [Result] Richards KC, Sullivan SC, Phillips RL, Beck CK, Overton-McCoy AL. The effect of individualized activities on the sleep of nursing home residents who are cognitively impaired: a pilot study. J Gerontol Nurs. 2001 Sep;27(9):30-7. doi: 10.3928/0098-9134-20010901-07. PMID 11820554
- [Result] Kolanowski AM, Richards KC, Sullivan SC. Derivation of an intervention for need-driven behavior. Activity preferences of persons with dementia. J Gerontol Nurs. 2002 Oct;28(10):12-5. doi: 10.3928/0098-9134-20021001-06. No abstract available. PMID 12382454
- [Result] Richards KC, Lambert C, Beck CK. Deriving interventions for challenging behaviors from the need-driven dementia-compromised behavior model. Alzheimer's care today. 2000 Oct 15; 1(4):62-76.